CLINICAL TRIAL: NCT00247429
Title: Vandral Retard (Venlafaxine Extended Release) in Depressive Syndrome With Anxiety and Painful Symptoms in Elderly Patients. Observational Study in Primary Care
Brief Title: Study Evaluating Venlafaxine Extended Release in Elderly Depressed Patients
Status: Completed | Type: Observational
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Other Study IDs: 101356
Record Dates: First submitted 2005-10-28; First posted 2005-11-01 (Estimated); Last update posted 2009-09-01 (Estimated); Status verified 2009-08

CONDITIONS: Depressive Syndrome; Anxiety
Keywords: depression; anxiety; elderly
MeSH Terms: conditions — Depressive Disorder; Anxiety Disorders; Depression

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: None Retained — No specimen retained

SUMMARY:
In this study we will assess as a primary objective the effect of venlafaxine retard treatment on primary care attended elderly patients with depressive syndrome. We will also study secondarily its effects on anxiety, somatic and painful symptoms of depression.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 60 years
* Depressive syndrome with associated anxiety symptoms, according to a symptoms intensity HAM-D17³14

Exclusion Criteria:

* Participation in other studies in the last 3 months before the start of the study
* Known hypersensibility to venlafaxine
* Clinically significant abnormalities according to the venlafaxine labeling

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary care centers
Sampling Method: Non-Probability Sample
Enrollment: 59 (Actual)
Dates: Start 2004-07; Primary Completion 2005-10 (Actual); Study Completion 2005-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Principal Investigator — Wyeth is now a wholly owned subsidiary of Pfizer